CLINICAL TRIAL: NCT01885065
Title: Efficacy Study of Novel Edible Gel-based Artificial Saliva in Xerostomic Cancer Patients
Brief Title: Efficacy of Novel Edible Gel-based Artificial Saliva in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dental Innovation Foundation Under Royal Patronage (Other)
Collaborators: Thammasat University (Other); Srinakharinwirot University (Other); Mahidol University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DIF-02
Record Dates: First submitted 2013-06-16; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Cancer of Head and Neck; Cancer; Radiation-induced Xerostomia; Dry Mouth
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gel-based artificial saliva (Experimental): Continuous oral intake of edible gel-based artificial saliva (30-50 ml/day) for four weeks
  Interventions: Other: Gel-based artificial saliva

INTERVENTIONS:
Other: Gel-based artificial saliva — Gel-based artificial saliva is an edible non-nutritious gel intended to relieve dry mouth.
  Taking orally 1-2 teaspoon each time, 5 times / day (30-50 ml/ day) for four weeks.
  Other Names: Oral moisturizing jelly

SUMMARY:
The purpose of this study is to determine whether continuous use of edible, gel-based artificial saliva in cancer patients with dry mouth problems will reduce signs and symptoms of dry mouth and improve quality of patients' saliva.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients who receive/ had received radiotherapy and/or chemotherapy and have dry mouth problems

Exclusion Criteria:

* mucositis more than grade 1
* cannot perform oral intake of gel-based artificial saliva eg. aspirate

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in subjective dry mouth score | baseline, 2 weeks and 4 weeks after intervention
  The outcome measure (subjective dry mouth score) will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)

SECONDARY OUTCOMES:
Changes in objective dry mouth score | Baseline, 2 week and 4 weeks after the start date
  The outcome measure will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)
Changes in salivary pH | Baseline, 2 weeks and 4 weeks after the start date
  The outcome measure will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)
Changes in salivary buffering capacity | Baseline, 2 weeks and 4 weeks after the start date
  The outcome measure will be measured before and 2 and 4 weeks after continuous usage of edible gel-based artificial saliva (30-50 ml/day for at least 5 days per week)

CONTACTS AND LOCATIONS:
Overall Officials: Aroonwan Lam-ubol, DDS, PhD, Study Chair — Faculty of Dentistry, Srinakharinwirot University
Locations (1):
- Mahavachiralongkorn cancer hospital, Pathum Thani, Changwat Pathum Thani, Thailand

REFERENCES:
- See also: Dental Innovation Foundation under Royal Patronage, His Majesty the King's Dental Service Unit — http://www.dent-in-found.org/